CLINICAL TRIAL: NCT06026514
Title: A Phase I Study of the Safety and Immunogenicity of the Recombinant, Live-Attenuated, Bovine/Human Parainfluenza Virus Vector Vaccine Expressing the 6P-Prefusion-Stabilized Version of the SARS-CoV-2 Spike Protein, Administered in Two Sequential Doses as Nasal Spray to Adults 18 to 50 Years of Age
Brief Title: Phase I Safety Study of B/HPIV3/S-6P Vaccine Via Nasal Spray in Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Johns Hopkins Bloomberg School of Public Health (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: CIR 355
Record Dates: First submitted 2023-08-30; First posted 2023-09-07 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: SARS-CoV-2 Infection
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Recombinant, Live-Attenuated, Bovine/Human Parainfluenza Virus Vector Vaccine Expressing the 6P-Prefusion-Stabilized Version of the SARS-CoV-2 Spike Protein, Administered in two Sequential Doses as Nasal Spray to Adults 18 to 50 Years of Age
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Intranasal Vaccine (Experimental): B/HPIV3/S-6P vaccine intranasally given in 2 doses, 56 days apart.
  Interventions: Biological: B/HPIV3/S-6P

INTERVENTIONS:
Biological: B/HPIV3/S-6P — Intranasal vaccine.

SUMMARY:
This Phase 1 clinical trial will evaluate the safety and immunogenicity of an intranasal vaccine candidate, a recombinant, live-attenuated, bovine/human parainfluenza virus vector vaccine expressing the 6-P prefusion-stabilized version of the SARS-CoV-2 spike protein.

DETAILED DESCRIPTION:
The proposed study is a single center, open label study to be conducted at the Johns Hopkins Bloomberg School of Public Health, Center for Immunization Research (CIR) in Baltimore, MD. Participants will be followed for 12 months after the first immunization, so the duration of study participation will be 12 months after receipt of initial vaccination.

Approximately 30 subjects will be enrolled in a rolling fashion to receive 2 doses of the B/HPIV3/S-6P vaccine intranasally 56 days apart. Participants who are enrolled and receive the first vaccine dose will not be replaced, even in the event they are ineligible or unable to take the second dose.

Up to 60 subjects will be consented to ensure that 30 subjects are eligible for enrollment and vaccination. Volunteers will be enrolled in a staggered fashion:

Group 1: Up to 5 volunteers will be enrolled and vaccinated. Group 2: Up to 10 volunteers will be enrolled and vaccinated. Group 3: The remaining volunteers (up to 15) will be enrolled and vaccinated.

ELIGIBILITY:
Inclusion Criteria:

1. Nonpregnant adults between 18 years and 50 years of age, inclusive.
2. General good health, without significant medical illness, physical examination findings, or significant laboratory abnormalities as determined by the investigator.
3. Demonstrates comprehension of the protocol procedures and knowledge of the trial by passing a written comprehension examination (passing grade > 70%).
4. Available for the duration of the trial.
5. Willingness to participate in the study and cooperate with the study procedures as evidenced by signing the informed consent document.
6. Persons of childbearing potential must have used effective birth control methods for at least one month prior to vaccination, and agree to continue with 'per label/fully effective use' for the chosen method for the duration of the study (30 days prior to first vaccination until 12 months after first vaccination), from amongst these:

   * pharmacologic/hormonal contraceptives, including oral, parenteral, subcutaneous, and transcutaneous delivery;
   * condoms or diaphragm with spermicide;
   * intrauterine device;
   * absolute abstinence from heterosexual intercourse as a matter of normal preferred lifestyle;
   * or must be surgically sterile or have documented menopause, having had no menses at all for at least one full year.

   All persons of childbearing potential must provide samples for urine and serum pregnancy testing prior to enrollment and prior to vaccination. Pregnancy risk assessment and pregnancy prevention counseling will occur at each point of contact.
7. Willingness to refrain from blood donation during participation in the study and for at least 1 year after receiving the second dose of vaccine.
8. Willingness to refrain from receiving vaccines or other investigational products during the first 90 days of the study after enrollment.

Exclusion Criteria:

1. Pregnancy as determined by a positive human choriogonadotropin (ßHCG) test in a person of reproductive capacity.
2. Currently breastfeeding.
3. Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, or renal disease by history, physical examination, electrocardiogram (EKG), and/or laboratory studies.
4. Behavioral or cognitive impairment or psychiatric disease that in the opinion of the investigator affects the ability of the subject to understand and cooperate with the study protocol.
5. A history of asthma within the past 5 years, or a current diagnosis of asthma or reactive airway disease associated with exercise, seasonal hay fever or allergic rhinitis.
6. Presence of any febrile illness or symptoms suggestive of a respiratory infection within 2 weeks prior to inoculation.
7. Use of systemic or nasal steroid preparations or immunosuppressive drugs within 30 days prior to vaccination. Topical steroid preparations are permitted.
8. Inhaled bronchodilator or inhaled steroid use within the last year or use after upper respiratory tract infections within the last 5 years.
9. Current or past (in the last 4 weeks) use of intranasal medications (including steroids, decongestants, or hormonal medications), or planning to use them within 28 days of study vaccination.
10. Evidence of current alcohol or illicit drug abuse or addiction.
11. Other condition that in the opinion of the investigator would jeopardize the safety or rights of a subject participating in the trial or would render the subject unable to comply with the protocol.
12. Positive ELISA and confirmatory tests for human immunodeficiency virus (HIV).
13. Positive ELISA and confirmatory test (e.g., recombinant immunoblot assay) for hepatitis C virus (HCV).
14. Positive hepatitis B virus surface antigen (HBsAg) by ELISA.
15. Known immunodeficiency syndrome.
16. Receipt of a live vaccine within 4 weeks or a killed vaccine within 2 weeks prior to receipt of the study vaccine or planned receipt within 90 days after vaccination. (Exception, influenza vaccine may be obtained more than 2 weeks after or prior to the study vaccine).
17. History of a surgical splenectomy.
18. Receipt of blood or blood-derived products (including immunoglobulin [Ig]) within 6 months prior to study inoculation.
19. Has participated in another investigational study involving any investigational product within 30 days, or 5 half-lives, whichever is longer, before the first vaccine administration.
20. Body mass index (BMI) < 18.5 or >40.
21. Any significant abnormality of the nose or nasopharynx, including recurrent epistaxis and including nasal or sinus surgery.
22. History of Bell's palsy.
23. Has a confirmed SARS-CoV-2 infection or COVID-19 vaccine/booster within 16 weeks prior to enrollment.
24. Unwillingness to have nasopharyngeal (NP) or blood samples saved for future respiratory virus research.
25. Pulmonary function test (PFT) testing for FVC, FEV1, FEV1% and PEF of <80 or incentive spirometer value < normal parameters based on gender, age, and height.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2023-09-18 (Actual); Primary Completion 2025-01-16 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
To determine the frequency of vaccine-related solicited adverse events (AEs) | During study days 0 to 28 and 56 to 84 (28 days after each dose)
  Summary and line listing of individual clinical solicited of the frequency of solicited AEs
To determine the frequency of vaccine-related unsolicited AEs | During study days 0 to 28 and 56 to 84 (28 days after each dose)
  Summary and line listing of individual clinical solicited of the frequency of unsolicited AEs
To determine the frequency of vaccine-related lower respiratory illness | During study days 0 to 28 and 56 to 84 (28 days after each dose)
  Summary and line listing of individual clinical solicited of the frequency of vaccine-related lower respiratory illness
Vaccine virus shedding on 1 or more days | On Days 4, 7, and 10, and 60, 63, and 66
  As assessed by culture, or rRT-PCR
Evidence of a >4-fold rise in HPIV3 antibody titers | When comparing pre-vaccination titers day 29, 56 or 90
  Using PRNT60 or ELISA

SECONDARY OUTCOMES:
Rise in serum neutralizing antibody titer to SARS-CoV-2 S protein | On days 63, 70, 84, 180, 360
  Will be measured by ELISA and neutralization assay

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland, United States